CLINICAL TRIAL: NCT04753398
Title: One Heart to Care for, Your Heart to Take Care of.
Brief Title: One Heart to Care for
Acronym: 1H2C4
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients included
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other); WGK Limburg (Unknown)
Responsible Party: Principal Investigator, Pieter Vandervoort, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 13/085U
Record Dates: First submitted 2014-03-03; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Telemonitoring; medication up titration; automatic blood pressure device; medication dispenser
MeSH Terms: conditions — Heart Failure | interventions — Blood Pressure Monitors

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemonitoring group (Experimental): Additional telemonitoring devices: Blood Pressure Monitor, medication dispenser, telemonitoring technology
  Interventions: Device: Blood Pressure Monitor, medication dispenser, telemonitoring technology
- Control group (No Intervention): usual care, without telemonitoring

INTERVENTIONS:
Device: Blood Pressure Monitor, medication dispenser, telemonitoring technology — The telemonitoring interference in the telemonitoring arm consists of an automatic blood pressure device and medication dispenser that transmit data to a central platform.
  Other Names: Telemedicine; remote monitoring; remote follow-up
  Arms: Telemonitoring group

SUMMARY:
This is an open randomized clinical trial with two study arms. One group, receiving usual care for heart failure, will be compared to another group, receiving usual care plus active telemonitoring interference.

When leaving the hospital, the usual care arm receives a document with a predefined medication scheme and advice for the general practitioner (like it is currently done in usual care). Besides the normal consultations at 2 and 5 weeks, no active interactions take place between the study nurse and the patient.

The telemonitoring interference in the other study arm consists of an automatic blood pressure device and medication dispenser that transmit data to a central platform. During the first 12 weeks, the nurse of the call center will give incentive for medication up titration on the basis of the available data. Before up titration can be done, the patient needs to take blood pressure measurements 3 times in the morning and 3 times in the evening and at least 6 measurements a week.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 50
* Patient has to be followed in Ziekenhuis Oost-Limburg or Jessa Ziekenhuis Hasselt
* The patient has to be able to live independently or in a service flat
* The diagnosis of heart failure or severe myocardial infarction has to be done after September 1, 2013 according to:

  * Left ventricular ejection fraction (LVEF) <40%
  * eGFR>30ml/min/kg
  * Treatment minimally with ACE-I and BB
* The general practitioner had to give his approval for the installation of telemonitoring On the basis of an interview between the heart failure nurse and patient, one will decide if the patient is eligibil to join the study. The patient also needs to speak sufficient Dutch to be communicative about his/her medical condition.

Exclusion Criteria:

* Reversible form of heart failure
* Heart failure due to severe aortic stenosis
* eGFR less than 30ml/min/kg
* Presence of a cardiac resynchronization therapy (CRT) device
* Palliative status following the RIZIV guidelines or according to the assessment of the cardiologist (<1 year)
* Patients staying in a nursing or retirement home
* Active treatment with either ACE-I/ARB or BB

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mean medication doses | week 12
  Define whether the mean medication doses of angiotensin-converting-enzyme inhibitor (ACE-I) and bètablockers (BB) in the group with telemonitoring is higher than in the group with usual care (without telemonitoring) after 12 weeks.
Mean medication doses | week 24
  Define whether the mean medication doses of angiotensin-converting-enzyme inhibitor (ACE-I) and bètablockers (BB) in the group with telemonitoring is higher than in the group with usual care (without telemonitoring) after 6 months

SECONDARY OUTCOMES:
Medication titration | up to one year
  Mean doses ACE-I/angiotensin receptor blockers (ARB) en BB after 6 months
All-cause mortality | Up to one year
  All-cause mortality
All cardio-related hospitalisations (number and time) | Up to one year
  * Arrythmogenic nature
  * Ischemic nature
  * Heart failure nature
  * Valvular/surgical nature
  * Elektrofysiological nature (implantation ICD, CRT,…)
All heart failure hospitalisations | Up to one year
  * Treatment with (whether or not intravenous) diuretic therapy
  * Treatment with hemodynamic guided therapy (vasodilators)
  * Treatment with intravenous inotropics
Number of medical practitioner-patient contacts | Up to one year
  * In hospital (medical record)
  * At patient home (WGK)
Number of (telephone) contacts, registered by the heart failure nurse | Up to one year
  Number of (telephone) contacts, registered by the heart failure nurse
Number of (telephone) contacts for the encouragement of medication compliance | Up to one year
  Number of (telephone) contacts for the encouragement of medication compliance
Evolution of heart failure and comorbidities | up to one year
  * Blood collection with: kidney function determinations, electrolytes, heart markers (NT-proBNP)
  * Echo parameters (cardiac output, LVEF, diameters end systolic and diastolic)
  * Exercise stress tests (VO2max, maximal wattage, maximal heart rate)
  * Weight, length, blood pressure, ECG
Quality of life according to the HeartQoL questionnaire | day 1, month 12
Satisfaction survey | month 12
  Satisfaction survey about the received care (anonymous)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Vandervoort, prof. dr., Principal Investigator — Ziekenhuis Oost-Limburg; Brenda Aendekerk, MSc, Study Director — Wit Gele Kruis Limburg, Genk, Belgium; Valerie Storms, dr., Study Director — Hasselt University; Lars Grieten, dr., Principal Investigator — Hasselt University; Christophe Smeets, MSc, Study Chair — Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium